CLINICAL TRIAL: NCT01272570
Title: Oral Health and Oral Health-Related Quality of Life in Early Stage Breast Cancer Survivors: The Role of Aromatase Inhibitors
Brief Title: Oral Health and Oral Health-Related Quality of Life in Early Stage Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Linda Susan Taichman, Assistant Professor of Dentistry, University of Michigan
Other Study IDs: HUM00036200
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer; Xerostomia
Keywords: breast; oral; cancer
MeSH Terms: conditions — Breast Neoplasms; Xerostomia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aromatase Inhibitor: * Diagnosis of BCa- Histologic confirmed diagnosis of BCa: Stage 0, I, II, or III with no evidence of metastatic disease.
  * Treatment- AI as clinically indicated (AI may be anastrozole, exemestane or letrozole). Subjects may have had prior tamoxifen or raloxifene. Subjects may have had chemotherapy and/or radiation therapy. Must be within the first year of consecutive AI therapy. If a subject started AI, discontinued, then restarted, they will be accepted into the study as long as the past therapy did not exceed 12 months and the current therapy has not exceeded 12 months.
- Control: • No Diagnosis of cancer.- Patients must not have a diagnosis of any cancer (Not including a history of thyroid or skin cancer).

SUMMARY:
The 3 Specific Aims are (1) To determine the prevalence, incidence and severity of oral conditions in postmenopausal early stage breast cancer survivors within the first 18 months of adjuvant Aromatase Inhibitor(AI) therapy, (2) To determine the oral health quality of life among postmenopausal early stage breast cancer survivors who are receiving AI therapy, (3) To determine the utilization of dental care among postmenopausal women receiving AIs with a history of early stage BCa over time. The hypothesis for this pilot study is that AIs negatively impact oral health and oral health quality of life in the setting of breast cancer survivors. Further, we hypothesize that dental visits are underutilized in women with BCa undergoing adjuvant AI therapy.

DETAILED DESCRIPTION:
This is a 2 arm prospective study. PM women receiving breast care, with and without breast cancer, at the University of Michigan are eligible. The study procedures include: survey/questionnaires, oral exam performed at Michigan Center for Oral Health Research (MCOHR) with specimen collection, and medical chart review. The goal of this study is to collect dental data and oral health quality of life data on women who are receiving AI therapy. This study does not administer any treatments or drugs to participants.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal as defined by NCCN (any of the following)

  * Prior bilateral oophorectomy
  * Age equal to or greater then 60 years of age
  * Age less then 60 and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression and FSH and estradiol in the postmenopausal range
  * If taking tamoxifen or toremifene and age less then 60y, then FSH and plasma estradiol level in postmenopausal ranges71.
* Individuals capable of consenting and self administering the survey instrument.
* At least 15 teeth present.

AI users:

* Diagnosis of BCa- Histologic confirmed diagnosis of BCa: Stage 0, I, II, or III with no evidence of metastatic disease.
* Treatment- AI as clinically indicated (AI may be anastrozole, exemestane or letrozole). Subjects may have had prior tamoxifen or raloxifene. Subjects may have had chemotherapy and/or radiation therapy. Must be within the first year of consecutive AI therapy. If a subject started AI, discontinued, then restarted, they will be accepted into the study as long as the past therapy did not exceed 12 months and the current therapy has not exceeded 12 months.

Controls:

-No Diagnosis of cancer.- Patients must not have a diagnosis of any cancer (Not including a history of thyroid or skin cancer).

Exclusion Criteria:

* Metastatic BCa (AI treated group: fully resected locally recurrent disease is permitted if the patient has been rendered without evidence of disease).
* Significant psychiatric illness/social situations that would preclude completion of questionnaires
* Chronic medications known to affect the periodontal status (calcium antagonist, anti-convulsives, immunosuppressives (> prednisone 7.5mg daily). NSAIDS and bisphosphonates are permitted.
* Premedication- Conditions that require antibiotic therapy will be evaluated on a case-by-case basis. (Patients taking prophylaxis for joint replacements will not be excluded.)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 29 postmenopausal women with a history of early stage BCa receiving adjuvant AI therapy and 29 postmenopausal women without cancer
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Periodontal diseases | At the time of study visit

SECONDARY OUTCOMES:
Oral health quality of life | At the time of study visit

CONTACTS AND LOCATIONS:
Overall Officials: Linda (Susan) Taichman, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Ries LA YJ, Keel GE, Eisner MP, Lin YD, Horner MJ. SEER Survival Monograph: Cancer Survival Among Adults: U.S. SEER Program, 1988-2001, Patient and Tumor Characteristics. . , Bethesda, MD,: National Cancer Institute, SEER Program, ; 2007.
- [Background] Sonis ST, Fey EG. Oral complications of cancer therapy. Oncology (Williston Park). 2002 May;16(5):680-6; discussion 686, 691-2, 695. PMID 12108892
- [Background] Stokman MA, Sonis ST, Dijkstra PU, Burgerhof JG, Spijkervet FK. Assessment of oral mucositis in clinical trials: impact of training on evaluators in a multi-centre trial. Eur J Cancer. 2005 Aug;41(12):1735-8. doi: 10.1016/j.ejca.2005.04.030. PMID 16039109
- [Background] Ohrn KE, Wahlin YB, Sjoden PO. Oral status during radiotherapy and chemotherapy: a descriptive study of patient experiences and the occurrence of oral complications. Support Care Cancer. 2001 Jun;9(4):247-57. doi: 10.1007/s005200000214. PMID 11430420
- [Background] Anderson WF, Chatterjee N, Ershler WB, Brawley OW. Estrogen receptor breast cancer phenotypes in the Surveillance, Epidemiology, and End Results database. Breast Cancer Res Treat. 2002 Nov;76(1):27-36. doi: 10.1023/a:1020299707510. PMID 12408373
- [Derived] Taichman LS, Van Poznak CH, Inglehart MR. Self-reported oral health and quality of life of postmenopausal breast cancer survivors on aromatase inhibitors and women without cancer diagnoses: a longitudinal analysis. Support Care Cancer. 2016 Nov;24(11):4815-24. doi: 10.1007/s00520-016-3336-6. Epub 2016 Jul 25. PMID 27455851